CLINICAL TRIAL: NCT00004156
Title: Vaccination of High Risk Breast Cancer Patients With MUC-1 (Glycosylated) Keyhole Limpet Hemocyanin Conjugates Plus the Immunological Adjuvant QS21
Brief Title: Vaccine Therapy in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-023; CDR0000067394 (Registry Identifier: PDQ (Physician Data Query)); NCI-H99-0043
Record Dates: First submitted 1999-12-10; First posted 2004-05-20 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- Vaccine: MUC1-KLH vaccine/QS21 (Experimental): Patients receive glycosylated MUC-1 antigen containing MUC-1(106) or MUC-1(33) with keyhole limpet hemocyanin conjugate subcutaneously (SQ) plus immunological adjuvant QS21 SQ on weeks 1-3, 7, and 19 for a total of 5 vaccinations. Patients are followed every 3 months.
  Interventions: Biological: MUC1-KLH vaccine/QS21

INTERVENTIONS:
Biological: MUC1-KLH vaccine/QS21

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine if immunization with glycosylated MUC-1 antigen containing MUC-1(106) or MUC-1(33) with keyhole limpet hemocyanin conjugate plus immunological adjuvant QS21 induces an antibody, helper T cell and/or cytotoxic T cell response against MUC-1 in patients with high risk breast cancer expressing MUC-1.

OUTLINE: Patients receive glycosylated MUC-1 antigen containing MUC-1(106) or MUC-1(33) with keyhole limpet hemocyanin conjugate subcutaneously (SQ) plus immunological adjuvant QS21 SQ on weeks 1-3, 7, and 19 for a total of 5 vaccinations. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosed breast cancer at high risk for disease recurrence with one of the following requirements: Disease free stage IV breast cancer following eradication of disease by surgery, radiotherapy, or chemotherapy Stage I, II, or III breast cancer remaining clinically free of identifiable disease following adjuvant chemotherapy with 2 consecutively rising CA15.3 (BR2729) or CEA levels at least 2 weeks apart Elevation of marker levels not needed for stage III disease if adjuvant therapy completed within past 2 years CEA increase at least 1.5 times upper chronic value in patients with significant smoking history and chronic CEA elevation less than 15 Recurrence in the ipsilateral axilla following lumpectomy/axillary dissection or modified radical mastectomy Recurrence in the ipsilateral breast following lumpectomy/axillary dissection Stage II disease with at least 4 positive axillary lymph nodes and adjuvant therapy completed within past 2 years Stable stage IV disease on hormonal therapy Colonoscopy required for isolated CEA elevation Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: Karnofsky 90-100% Life expectancy: Not specified Hematopoietic: Lymphocyte count at least 500/mm3 WBC at least 3,000/mm3 Hepatic: Alkaline phosphatase no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 1.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No New York Heart Association class III or IV heart disease Other: No immunodeficiency or autoimmune disease No seafood allergies No other active malignancies except basal cell or squamous cell skin cancer Not pregnant Negative pregnancy test Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 weeks since prior immunotherapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy No concurrent chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy No concurrent radiotherapy Surgery: See Disease Characteristics At least 4 weeks since prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1999-05; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
immune response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Ann Gilewski, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Musselli C, Ragupathi G, Gilewski T, Panageas KS, Spinat Y, Livingston PO. Reevaluation of the cellular immune response in breast cancer patients vaccinated with MUC1. Int J Cancer. 2002 Feb 10;97(5):660-7. doi: 10.1002/ijc.10081. PMID 11807794